CLINICAL TRIAL: NCT05842694
Title: Mid-Term Outcomes Of Fracture Odontoid Management in Assiut University
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Osama Mohamed Emam, principal investigator, Assiut University
Other Study IDs: follow up of Odontoid fracture
Record Dates: First submitted 2023-03-31; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Cervical Spine Fracture

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to evaluate and assess the mid-term outcomes of treating odontoid fracture cases admitted to the Trauma Unit of Assiut University Hospital.

DETAILED DESCRIPTION:
Odontoid fractures are common fractures of the cervical spine, accounting for 10-15% of all cervical spine fractures. It has a bimodal age distribution as it occurs in both elderly and young patients. The injury generally occurs as a result of strong flexion and extension movement in addition to axial overload. Flexion generally results in anterior subluxation, while extension results in posterior subluxation.

It was classified by Anderson and D'Alonzo Classification in 1974 into three types according to the fracture location. A newer classification was introduced which offered a clearer distinction between type-II and type-III fractures. In this new classification, Type II fractures were further divided into 3 subtypes. The 3 subtypes are labelled A, B, and C. Type II fractures are usually treated surgically through either anterior or posterior approach depending on the fracture pattern as they are characterized by a higher rate of non-union compared to type I and III being in a watershed level between the vertebral and the internal carotid arteries. Nevertheless, the literature is still confusing about the results of anterior surgery in odontoid fractures.

In a recent study by Cutler et al., anterior fixation of odontoid fracture was associated with high morbidity and mortality. In another study, the most commonly reported major complications after odontoid fracture surgery in the elderly include cardiac failure, deep venous thrombosis , stroke, pneumonia, respiratory failure, liver failure, and severe infection.

Despite the fact that we receive and treat a large number of patients with various types of odontoid fractures in Assiut University Hospital, there is no consensus about the best treatment options and uncertainty about the mid and long term outcome of these treatments.

In this study, the investigators will assess the mid-term outcomes (minimum of one year) to all patients with odontoid fracture who are admitted to the Trauma Unit in Assiut University Hospital regardless the treatment type.

ELIGIBILITY:
Inclusion Criteria:

* All patients with odontoid fractures presenting to Assiut University Hospital - Department of Orthopaedic and Trauma Surgery who have completed a minimum of 1 year follow up regardless of age, mechanism of injury, neurological status or type of treatment applied

Exclusion Criteria:

* Patients who are not available for one year follow-up Patients who refuse to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with odontoid fractures presenting to Assiut University Hospital - Department of Orthopaedic and Trauma Surgery who have completed a minimum of 1 year follow up regardless of age, mechanism of injury, neurological status or type of treatment applied
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-05-10 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
follow up of patients with odontoid fracture using neck disability index | baseline
  Percentage of improvement in neck disability index following conservative and surgical treatment during the follow up visits

SECONDARY OUTCOMES:
rate of complication | baseline
  1. Fracture healing
  2. Incidence and rate of complications (e.g. non-union, post-operative infections, C1-2 Instability, etc…..) Return to work/activity of daily living

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt

REFERENCES:
- [Background] Julien TD, Frankel B, Traynelis VC, Ryken TC. Evidence-based analysis of odontoid fracture management. Neurosurg Focus. 2000 Jun 15;8(6):e1. doi: 10.3171/foc.2000.8.6.2. PMID 16859271
- [Background] Chi YL, Wang XY, Xu HZ, Lin Y, Huang QS, Mao FM, Ni WF, Wang S, Dai LY. Management of odontoid fractures with percutaneous anterior odontoid screw fixation. Eur Spine J. 2007 Aug;16(8):1157-64. doi: 10.1007/s00586-007-0331-0. Epub 2007 Mar 3. PMID 17334793
- [Background] Grauer JN, Shafi B, Hilibrand AS, Harrop JS, Kwon BK, Beiner JM, Albert TJ, Fehlings MG, Vaccaro AR. Proposal of a modified, treatment-oriented classification of odontoid fractures. Spine J. 2005 Mar-Apr;5(2):123-9. doi: 10.1016/j.spinee.2004.09.014. PMID 15749611
- [Background] Cutler HS, Guzman JZ, Lee NJ, Kothari P, Kim JS, Shin JI, Leven DM, Cho SK. Short-Term Complications of Anterior Fixation of Odontoid Fractures. Global Spine J. 2018 Feb;8(1):47-56. doi: 10.1177/2192568217698132. Epub 2017 May 16. PMID 29456915
- [Background] White AP, Hashimoto R, Norvell DC, Vaccaro AR. Morbidity and mortality related to odontoid fracture surgery in the elderly population. Spine (Phila Pa 1976). 2010 Apr 20;35(9 Suppl):S146-57. doi: 10.1097/BRS.0b013e3181d830a4. PMID 20407346
- [Background] Vernon H, Mior S. The Neck Disability Index: a study of reliability and validity. J Manipulative Physiol Ther. 1991 Sep;14(7):409-15. PMID 1834753